CLINICAL TRIAL: NCT06763289
Title: Comparison Between Multi-omics Models Including DNA Methylation in CfDNA, Quantitative Determination of Epstein-Barr Virus Nucleic Acid and Serological Double Antibody Detection in Early Screening of Nasopharyngeal Carcinoma
Brief Title: Comparison of Multi-omics Models for Early Nasopharyngeal Carcinoma Screening: CfDNA Methylation, EBV DNA, and Serological Double-antibodies Detection
Acronym: PROFOUND-NPC
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Hainan People's Hospital (Other); Xiangya Hospital of Central South University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Weiping Wen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PROFOUND-NPC
Record Dates: First submitted 2024-12-21; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: cell-free DNA; methylation; cancer early detection
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case arm: Participants with newly diagnosed cancer of nasopharyngeal carcinoma
- Control arm: Participants without a cancer diagnosis after routine cancer screening tests.

SUMMARY:
This study focus on nasopharyngeal carcinoma, a cancer type with Chinese characteristics, analyze the early screening detection performance of nasopharyngeal carcinoma in the multi-cancer early screening model, and compare the performance differences among multi-omics models such as nasopharyngeal carcinoma-specific DNA methylation and fragmentome in the multi-cancer early screening model and the clinically routinely conducted Epstein-Barr virus (EBV) nucleic acid quantification (EBV DNA) test and serological double antibody (double antibodies of EBNA1-IgA and VCA-IgA) test. It suggests that compared with EBV DNA quantification and double antibody tests, in patients with nasopharyngeal carcinoma, multi-omics models such as DNA methylation can avoid false negatives, improve sensitivity, and increase the detection rate of early-stage nasopharyngeal carcinoma; in patients without nasopharyngeal carcinoma, multi-omics models such as DNA methylation can avoid false positives, improve specificity, and avoid unnecessary over-diagnosis.

ELIGIBILITY:
Inclusion Criteria for Case Arm Participants:

1. 40-74 years old
2. Clinically and/or pathologically diagnosed cancer
3. No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
4. Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria for Case Arm Participants:

1. Pregnancy or lactating women
2. Known prior or current diagnosis of other types of malignancies comorbidities
3. Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
4. Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
5. Recipients of blood transfusion within 30 days prior to screen
6. Recipients of therapy in past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
7. Unsuitable for this trial determined by the researchers

Inclusion Criteria for Control Arm Participants:

1. 40-74 years old
2. Without confirmed cancer diagnosis
3. Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria for Control Arm Participants:

1. Pregnancy or lactating women
2. Known prior or current diagnosis of other types of malignancies comorbidities
3. Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
4. Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
5. Recipients of blood transfusion within 30 days prior to screen
6. Recipients of therapy in the past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
7. Unsuitable for this trial determined by the researchers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed cancers or individuals without confirmed cancer will be invited to participate in this case-control study by a designated consenting professional.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
False positive rate and false negative rate of ctDNA Methylation model, EBV DNA quantification test, double antibodies of EBNA1-IgA and VCA-IgA test | 2 year
  To analyze the early screening detection performance of nasopharyngeal carcinoma in the multi-cancer early screening model, and compare the false positive rate and false negative rate among in the multi-cancer early screening model and the clinically routinely conducted Epstein-Barr virus (EBV) nucleic acid quantification (EBV DNA) test and serological double antibody (double antibodies of EBNA1-IgA and VCA-IgA) test.
Sensitivity and specificity of ctDNA Methylation model, EBV DNA quantification test, double antibodies of EBNA1-IgA and VCA-IgA test in the Screening of nasopharyngeal carcinoma | 2 year
  To analyze the early screening detection performance of nasopharyngeal carcinoma in the multi-cancer early screening model, and compare the sensitivity and specificity among in the multi-cancer early screening model and the clinically routinely conducted Epstein-Barr virus (EBV) nucleic acid quantification (EBV DNA) test and serological double antibody (double antibodies of EBNA1-IgA and VCA-IgA) test.

SECONDARY OUTCOMES:
Sensitivity and specificity of ctDNA Methylation model, EBV DNA quantification test, double antibodies of EBNA1-IgA and VCA-IgA test in the detection of early-stage nasopharyngeal carcinoma | 2 year
  To analyze the early screening detection performance of nasopharyngeal carcinoma in the multi-cancer early screening model, and compare the sensitivity and specificity among in the multi-cancer early screening model and the clinically routinely conducted Epstein-Barr virus (EBV) nucleic acid quantification (EBV DNA) test and serological double antibody (double antibodies of EBNA1-IgA and VCA-IgA) test in the detection of stage I/II nasopharyngeal carcinoma.
Modeled positive and negative predictive values of ctDNA Methylation model, EBV DNA quantification test, double antibodies of EBNA1-IgA and VCA-IgA test | 2 year
  The difference in positive and negative predictive values was calculated combined with the incidence of nasopharyngeal carcinoma and compared among in the multi-cancer early screening model and the clinically routinely conducted Epstein-Barr virus (EBV) nucleic acid quantification (EBV DNA) test and serological double antibody (double antibodies of EBNA1-IgA and VCA-IgA) test.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No